CLINICAL TRIAL: NCT00611962
Title: Phase II Study of Combined Oxaliplatin and Paclitaxel for Metastatic Germ Cell Tumors
Brief Title: Phase II Study of Oxaliplatine-Paclitaxel in Patients With Metastatic Germ Cell Tumor Refractory to Cisplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Nathalie Billon/Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFC_7407
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-01

CONDITIONS: Neoplasms, Germ Cell and Embryonal
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Oxaliplatin; Paclitaxel

INTERVENTIONS:
Drug: Oxaliplatin, Paclitaxel — Oxaliplatin was provided in clear glass vials sealed with a rubber stopper and an aluminum seal with a flip-off cover. Each vial contained 50 or 100 mg of active ingredient with 450 or 900 mg, respectively, of lactose monohydrate as excipient
  Paclitaxel was supplied as single dose vials of 30 mg/5 mL or 100 mg/17 mL.
  Other Names: Eloxatin®, Taxol

SUMMARY:
To evaluate the efficacy of the oxaliplatin-paclitaxel combination i.e. evaluation of tumor response rate using World Health Organization/Union Internationale Contre le Cancer (WHO/UICC) and Indianapolis tumor marker (human chorionic gonadotropin [hCG], alpha fetoprotein [AFP]) criteria in metastatic germ cell cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven germ cell cancer: gonadal (including ovarian) or extragonadal, seminomatous or non seminomatous, or clinical presentation of a GCT with elevated AFP level and/or hCG level (> or =to 100 x ULN) when a biopsy was not available
* Metastatic GCT patients:
* Progression disease defined as > 10% increase in hCG and/or AFP markers (and/or documented progressive disease [PD]) during a platinum-based chemotherapy or less than 6 months after the last cycle (in the case of growing non seminomatous tumor, without increased markers, a histological documentation of malignant tumor was required, to exclude growing mature teratoma)
* At least 1 prior line of chemotherapy containing CDDP + etoposide; (prior regimen with high dose chemotherapy and hematopoietic stem cell support was permitted)
* Eastern Cooperative Oncology Group PS (ECOG PS) grade < or =to 2
* At least 1 bidimensionally measurable lesion by imaging (CT scan) of > or =to 20 mm outside an irradiated area OR significantly increased tumor markers > 2 x ULN (on > or =to 2 consecutive tests, even in the absence of measurable lesions)
* Age > or =to 18
* Adequate bone marrow reserve
* Neutrophil count > or =to 1500/mm3
* Platelets > or =to 100,000/mm3
* Renal function:Creatinine < 3 x ULN
* Liver function:Transaminases < or =to 2.5 x ULN, total bilirubin < 1.5 x ULN (if liver metastases, transaminases < or =to 5 x ULN)
* Laboratory values obtained in the week preceding study entry
* Neurosensory < or =to grade 1 NCI CTC
* Signed informed consent obtained prior to all study procedures

Exclusion Criteria:

* Concomitant high-dose steroids (except for antiemetic prophylaxis)
* Pregnancy, breast-feeding or absence of contraception in sexually active patients
* Prior treatment with oxaliplatin or taxanes
* History of second malignancy, except for cured non melanoma skin cancer or excised in situ cervical carcinoma
* Symptomatic cerebral and/or leptomeningeal metastasis (irradiated brain metastases not requiring corticosteroid treatment were allowed)
* Treatment with another experimental drug or anticancer agent or participation in another clinical study within 30 days prior to study
* Other serious illness or uncontrolled infection
* Psychological, social or geographical situation preventing regular follow-up
* Primary tumor in brain/central nervous system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2000-12; Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Evaluate efficacy of oxaliplatin-paclitaxel combination using established criteria in metastatic germ cell cancer patients | during the study conduct

SECONDARY OUTCOMES:
Evaluate safety, and toxicity using established criteria,specific neurotoxicity scales, serious adverse events (SAEs) and treatment withdrawals | During the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Billon, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Lyon, France